CLINICAL TRIAL: NCT02950259
Title: A Phase Ib Study to Assess the Safety, Tolerability and Immunologic Activity of Preoperative IRX 2 In Early Stage Breast Cancer
Brief Title: Pre-operative IRX-2 in Early Stage Breast Cancer (ESBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Brooklyn ImmunoTherapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-126B; IRX-2 2016-B (Other: IRX Therapeutics)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasm; Breast Neoplasm, Male; Triple Negative Breast Cancer
Keywords: Breast Cancer; Early Stage Breast Cancer; Male breast cancer; IRX-2; Immunotherapy; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; Indomethacin; Omeprazole; Geritol; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IRX-2 Regimen -Early Stage Breast Cancer (Experimental): Enrolled subjects with early stage breast cancer will receive a single dose of cyclophosphamide (300 mg/m2) by IV infusion on Day 1. Also starting on Day 1 and continuing until Day 21, subjects will take daily oral indomethacin (25 mg three times each day), daily oral omeprazole (one tablet) and daily oral multivitamin containing 15-30 mg of zinc. On any 10 consecutive day period between Days 4-17, patients will receive two 1 mL subcutaneous periareolar injections of IRX-2.
  Interventions: Drug: Cyclophosphamide; Drug: Indomethacin; Drug: Omeprazole; Dietary Supplement: Multivitamin
- IRX-2 Regimen -Triple Negative Breast Cancer (Experimental): Enrolled subjects with triple negative breast cancer will receive a single dose of cyclophosphamide (300 mg/m2) by IV infusion on Day 1. Also starting on Day 1 and continuing until Day 21, subjects will take daily oral indomethacin (25 mg three times each day), daily oral omeprazole (one tablet) and daily oral multivitamin containing 15-30 mg of zinc. On any 10 consecutive day period between Days 4-17, patients will receive two 1 mL subcutaneous periareolar injections of IRX-2.
  Interventions: Drug: Cyclophosphamide; Drug: Indomethacin; Drug: Omeprazole; Dietary Supplement: Multivitamin

INTERVENTIONS:
Drug: Cyclophosphamide — One dose of cyclophosphamide 300 mg/m2 IV infusion
  Other Names: Cytoxan
Drug: Indomethacin — Indomethacin 25 mg three times a day for 21 days
  Other Names: Indocin
Drug: Omeprazole — One tablet of omeprazole daily for 21 days
  Other Names: Prilosec
Dietary Supplement: Multivitamin — Daily multivitamin containing 15-30 mg of zinc for 21 days.
  Other Names: Vitamin

SUMMARY:
The goal of this study is assess the safety and tolerability of the IRX-2 regimen in patients with early stage breast cancer (ESBC) and to estimate the pathologic complete response rate to neoadjuvant anthracycline-based and non-platinum containing chemotherapy in patients with triple-negative breast cancer who have received the IRX-2 Regimen before chemotherapy.

DETAILED DESCRIPTION:
This will be a Phase Ib study conducted to determine the safety and tolerability of an IRX-2 regimen in ESBC, to be administered pre-operatively before standard-of-care surgical resection and following standard-of-care diagnostic biopsy. This study will also include triple-negative breast cancer patients who will receive the IRX-2 regimen prior to chemotherapy.

Eligible subjects will have early stage breast cancer of any receptor sub-type, for which standard-of-care surgical resection is planned. To be eligible, a minimum of 1 core of tumor-bearing biopsy material must be available for research analysis.

Cohort B will enroll subjects triple negative breast cancer (defined by ER<10%, PR<10%, and HER2-negative by NCCN guidelines), T1c+ tumors for which neoadjuvant anthracycline-based and non-platinum containing chemotherapy is planned. The IRX-2 regimen will be administered and completed preceding chemotherapy. Cohort B subjects must undergo post-IRX-2 Regimen biopsy (2-3 cores), followed by commencement of chemotherapy preferably within one week after biopsy.

The IRX-2 regimen will be administered in all enrolled subjects. IRX 2 will be administered by subcutaneous injection into the periareolar skin of the affected breast.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer of any receptor subtype diagnosed by core-needle biopsy
* To undergo surgical resection with curative intent by partial mastectomy (lumpectomy) or mastectomy or
* Triple negative breast cancer (defined by ER<10%, PR<10%, and HER2-negative by NCCN guidelines), T1c+ tumors for which neoadjuvant anthracycline-based and non-platinum containing chemotherapy is planned
* Tumor >5 mm in maximum diameter by ultrasound or mammography. (Subjects with smaller tumors may be included at the discretion of the Principal Investigator.)
* Willing and able to provide written informed consent, including consent for use of available tissue and required blood draws for research purposes
* Availability of at least one tumor-bearing core specimen from the breast cancer diagnostic biopsy
* Karnofsky Performance status (KPS) 70% or greater.
* Female or male ≥18 years of age on day of signing informed consent.
* Adequate organ function as defined by protocol specified lab results

Exclusion Criteria:

* Prior neoadjuvant systemic therapy is planned
* Prior surgery, radiotherapy or chemotherapy for this cancer (other than core-needle biopsy)
* Received an investigational agent within 4 weeks of the first dose of treatment.
* Diagnosis of immunodeficiency or has received more than replacement doses of corticosteroids any other immunosuppressive therapy within 4 weeks of the first dose of treatment
* Hypersensitivity to IRX 2, cyclophosphamide, indomethacin, aspirin or ciprofloxacin.
* Chronic anticoagulation, not including aspirin, but including heparins, warfarin, oral anticoagulants or other platelet function inhibitors, that cannot, in the documented opinion of the investigator, safely be interrupted from at least 2 days prior to the initiation of the study regimen until after surgical resection of the tumor.
* Another malignancy that required active treatment within 6 months of the first dose of treatment
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, such that trial participation is not in the best interest of the subject, including but not limited to uncontrolled hypertension or clinically significant cardiovascular disease, myocardial infarction within the previous 3 months, active infection or pneumonitis or other pulmonary disease requiring systemic therapy, clinically significant gastritis or peptic ulcer disease (that would preclude the use of indomethacin), stroke of other symptoms of cerebral vascular insufficient within the last 3 months, autoimmune disease that has required systemic treatment within the past 2 years (other than hormone replacement doses), or uncontrolled psychiatric or substance abuse disorders.
* Pregnancy or lactation.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2025-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Page, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Providence Health & Services has agreed to allow IRX Therapeutics to have access PHI for auditing purposes. Any non-Providence Health & Services employee who will access PHI will be required to sign a confidentiality agreement and will not be permitted to remove PHI from Providence Health & Services.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years
Access Criteria: IPD will be accessed for data verification purposes only.

REFERENCES:
- [Derived] Sanchez K, Kim I, Chun B, Pucilowska J, Redmond WL, Urba WJ, Martel M, Wu Y, Campbell M, Sun Z, Grunkemeier G, Chang SC, Bernard B, Page DB. Multiplex immunofluorescence to measure dynamic changes in tumor-infiltrating lymphocytes and PD-L1 in early-stage breast cancer. Breast Cancer Res. 2021 Jan 7;23(1):2. doi: 10.1186/s13058-020-01378-4. PMID 33413574
- See also: Providence Cancer Center — https://oregon.providence.org/our-services/p/providence-cancer-center/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to poor accrual, site opted against enrolling patients into cohort B in favor of a different trial which is ongoing.
Groups:
- Total: Total of all reporting groups
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer | Total
Number analyzed (Participants) | 16 | 0 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 12 |  | 12
  >=65 years | 4 |  | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 |  | 16
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 14 |  | 14
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 15 |  | 15
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 |  | 16
Menstrual Status [Count of Participants; unit: Participants]
  Premenopausal | 6 |  | 6
  Post-menopausal | 10 |  | 10
Family History of Breast/Ovarian Cancer [Count of Participants; unit: Participants]
  Yes | 5 |  | 5
  No | 10 |  | 10
  Unknown/Not Reported | 1 |  | 1
Known BRCA 1/2 Mutation [Count of Participants; unit: Participants]
  Yes | 3 |  | 3
  No | 1 |  | 1
  Unknown | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Establish the Safety of the IRX-2 Regimen When Administered Pre-operatively in Early Stage Breast Cancer (ESBC) Patients
Description: The safety of IRX-2 will be determined by any surgical delays associated with administration of the study regimen.
Time Frame: Day 1 to Day 26
Population: No patients were enrolled into Arm B due to poor accrual and opted against Arm B in favor of the NeoIRX trial.
Measure: Count of Participants; unit: Participants
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Number analyzed (Participants) | 16 | 0
Participants | 0 | 0

2. Secondary Outcome: Tumor Infiltrating Lymphocytes
Description: Change in tumor infiltrating lymphocyte (TIL) score as measured by hematoxylin and eosin tumor infiltrating lymphocytes (H&E TIL) count according to Salgado criteria from pre-surgical biopsy to resected tumor specimen
Time Frame: At time of pre-surgical biopsy and time of tumor specimen resection at day 26
Population: Due to poor patient accrual we opted against enrolling into Cohort B in favor of the neoIRX trial.
Measure: Median (Full Range); unit: percentage of stromal area
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Number analyzed (Participants) | 16 | 0
percentage of stromal area | 0.4 [-0.2 to 12.8] |

3. Other Pre Specified Outcome: Characterization of Peripheral Lymphocytes
Description: Fold change of peripheral lymphocytes including activated T-cells, T-regulatory cells, natural killer (NK) cells, and myeloid cells
Time Frame: Day 1 to Day 26
Population: Due to poor accrual we opted against enrolling in Cohort B in favor of the neoIRX trial.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Number analyzed (Participants) | 16 | 0
fold change
  Stroma, Any PD-L1: T-Cell (any type) | 2.01 [1.32 to 3.08] |
  Stroma, Any PD-L1: Helper T-Cell | 2.05 [1.14 to 3.70] |
  Stroma, Any PD-L1: Cytotoxic T-Cell | 2.55 [1.80 to 3.61] |
  Stroma, Any PD-L1: Regulatory T-Cell | 0.91 [0.60 to 1.39] |
  Stroma, Any PD-L1: Macrophage | 0.86 [0.54 to 1.38] |
  Stroma, PD-L1-positive: T-Cell (any type) | 3.54 [1.86 to 6.76] |
  Stroma, PD-L1-positive: Helper T-Cell | 3.58 [1.76 to 7.29] |
  Stroma, PD-L1-positive: Cytotoxic T-Cell | 2.98 [1.74 to 5.08] |
  Stroma, PD-L1-positive: Regulatory T-cell | 1.38 [0.78 to 2.46] |
  Stroma, PD-L1-positive: Macrophage | 1.63 [0.84 to 3.13] |
  Tumor, Any PD-L1: T-Cell (any type) | 1.07 [0.65 to 1.77] |
  Tumor, Any PD-L1: Helper T-Cell | 0.77 [0.49 to 1.22] |
  Tumor, Any PD-L1: Cytotoxic T-Cell | 1.36 [0.91 to 2.05] |
  Tumor, Any PD-L1: Regulatory T-Cell | 0.79 [0.49 to 1.29] |
  Tumor, Any PD-L1: Macrophage | 0.65 [0.38 to 1.09] |
  Tumor, PD-L1-positive: T-Cell (any type) | 1.50 [0.86 to 2.63] |
  Tumor, PD-L1-positive: Helper T-cell | 1.07 [0.56 to 2.04] |
  Tumor, PD-L1-positive: Cytotoxic T-Cell | 1.68 [1.06 to 2.64] |
  Tumor, PD-L1-positive: Regulatory T-Cell | 0.64 [0.32 to 1.29] |
  Tumor, PD-L1-positive: Macrophage | 0.87 [0.51 to 1.49] |
  Stoma and tumor, PD-L1-positive: PD-L1+ IC^3 | 3.14 [1.68 to 5.87] |

4. Other Pre Specified Outcome: TIL Phenotype
Description: Post-IRX mean density of T-regulatory cells, activated T-cells, myeloid lineages and dendritic cells post-IRX within stromal tissue compartments.
Time Frame: Day 1 to 26
Population: Due to poor patient accrual we opted against enrolling into Cohort B in favor of the neoIRX trial.
Measure: Mean (Standard Deviation); unit: count/pixel
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Number analyzed (Participants) | 16 | 0
count/pixel
  Any PD-L1: T-cell (any type) | 1.27 (0.15) |
  Any PD-L1: Helper T-cell | 0.79 (.59) |
  Any PD-L1: Cytotoxic T-cell | 0.42 (0.30) |
  Any PD-L1: Regulatory T-cell | 0.07 (0.06) |
  Any PD-L1: Macrophage | 0.19 (0.12) |
  PD-L1-positive: T-cell (any type) | 0.7 (0.59) |
  PD-L1-positive: Helper T-Cell | 0.47 (0.46) |
  PD-L1-positive: Cytotoxic T-Cell | 0.19 (0.21) |
  PD-L1-positive: Regulatory T-Cell | 0.05 (0.05) |
  PD-L1-positive: Macrophage | 0.14 (0.11) |

5. Other Pre Specified Outcome: Intratumoral T-cell Clonality Response
Description: Change in T-cell clonal responses by T-cell receptor DNA deep sequencing
Time Frame: Day 1-26
Population: Due to poor patient accrual we opted against enrolling into Cohort B in favor of the neoIRX trial.
Measure: Number; unit: fold change
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Number analyzed (Participants) | 16 | 0
fold change
  Patient 1 | 0.7 |
  Patient 2 | -0.2 |
  Patient 3 | -0.3 |
  Patient 4 | 0.00 |
  Patient 5 | 0.2 |
  Patient 6 | 0.0 |
  Patient 7 | 0.1 |
  Patient 8 | 0.2 |
  Patient 9 | -0.3 |
  Patient 10 | 0.2 |
  Patient 11 | 0.1 |
  Patient 12 | -0.1 |
  Patient 13 | -0.1 |
  Patient 14 | NA — Patient did not have available paired lymph node specimen available for analyzation. |
  Patient 15 | -0.2 |
  Patient 16 | 1.5 |

6. Other Pre Specified Outcome: Intratumoral Immune Response
Description: The Nanostring PanCancer Immune panel was used to estimate increase in PD-L1 mRNA expression among tumor-bearing FFPE specimens.
Time Frame: Day 1-26
Population: Due to poor patient accrual we opted against enrolling into Cohort B in favor of the neoIRX trial.
Measure: Number; unit: fold change
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
Number analyzed (Participants) | 16 | 0
fold change
  Patient 1 | .9 |
  Patient 2 | .6 |
  Patient 3 | 0 |
  Patient 4 | .7 |
  Patient 5 | 0 |
  Patient 6 | 0 |
  Patient 7 | .5 |
  Patient 8 | -.5 |
  Patient 9 | .5 |
  Patient 10 | 1.5 |
  Patient 11 | 1.8 |
  Patient 12 | 0 |
  Patient 13 | 0 |
  Patient 14 | 0 |
  Patient 15 | 1.6 |
  Patient 16 | .7 |

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Description: Adverse event monitoring/recording happened at set time intervals as per study protocol
Arm/Group | IRX-2 Regimen -Early Stage Breast Cancer | IRX-2 Regimen -Triple Negative Breast Cancer
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/0
Other Adverse Events (participants affected / at risk) | 16/16 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IRX-2 Regimen -Early Stage Breast Cancer (N=16) | IRX-2 Regimen -Triple Negative Breast Cancer (N=0)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bruising/Bruising at Injection Site (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flu-like Symptoms (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Intermittent Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left Axillary Lymph Node Pain (General disorders) | 1 (1) | 0 (0)
Left Breast Pain (General disorders) | 1 (1) | 0 (0)
Mild Pain with Injections (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 0 (0)
Pain with Injections (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT02950259/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02950259/ICF_001.pdf